CLINICAL TRIAL: NCT05556863
Title: A Randomized, Double-blind, Placebo-controlled Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ELA026 Following Intravenous and/or Subcutaneous Administration of Single and Multiple Doses in Healthy Adults
Brief Title: Evaluation of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ELA026 in Single and Multiple Doses in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Electra Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Other
Other Study IDs: ELA026-CP001
Record Dates: First submitted 2022-09-20; First posted 2022-09-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2023-10

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Single Ascending Dose (Experimental): Cohort 1 Single dose: 0.001 mg/kg IV
  Cohorts 2 - 11 Single dose: dose level and route (IV or SC) to be determined
  Japanese Cohort Single dose: dose level and route (IV or SC) to be determined
  Interventions: Drug: ELA026
- Part 2: Multiple Ascending Dose (Experimental): Cohort 1 - 6 Multi-dose: dose level, route (IV or SC) and frequency to be determined
  Interventions: Drug: ELA026

INTERVENTIONS:
Drug: ELA026 — Single dose of ELA026
  Arms: Part 1: Single Ascending Dose
Drug: ELA026 — Multiple doses of ELA026
  Arms: Part 2: Multiple Ascending Dose

SUMMARY:
ELA026 is a fully human IgG1 SIRP-directed monoclonal antibody designed to reduce the myeloid and T cells driving the inflammation. The purpose of this study is to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of ELA026 in Single and Multiple Doses in Healthy Adults.

DETAILED DESCRIPTION:
This is a multi-center, Phase 1, randomized, double-blind, placebo-controlled study to assess the safety, tolerability, PK, and PD of ELA026 following single and multiple IV and/or SC dose administration in healthy adult volunteers, including a subgroup of Japanese volunteers.

The study will consist of 2 parts:

* Part 1: single ascending doses (SAD) in up to 11 SAD cohorts plus a Japanese cohort
* Part 2: multiple doses (MD) up to 6 MD cohorts

ELIGIBILITY:
Inclusion Criteria:

1. Non-Japanese subjects 19 to 60 years of age. Japanese subjects 20 to 60 years of age.
2. Must be in good general health.
3. No clinically significant abnormal laboratory values during screening.
4. Body mass index of 18 - 32 kg/m2.

Exclusion Criteria:

1. Clinical diagnosis or laboratory evidence of renal, hepatic, central nervous system, respiratory, cardiovascular, or metabolic disease at Screening.
2. Diagnosed with any form of malignancy (except basal cell carcinoma, fully removed).
3. Clinically significant immunodeficiency or autoimmunity assessed by medical history and/or laboratory test results.
4. Active or latent tuberculosis (TB), regardless of treatment history,
5. Positive drug abuse test.
6. Positive HIV, HBV, HCV test results.
7. Clinically significant ECG test results.
8. Clinically significant vital sign results.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of Treatment-Emergent Adverse Events [Safety and Tolerability]. | By week 3

SECONDARY OUTCOMES:
Plasma concentrations of ELA026 | By week 3
Change from baseline of monocytes levels. | By week 3
Change from baseline of lymphocytes levels. | By week 3
Presence of Anti-drug antibodies to ELA026 | By week 3
Comparison of ELA026 Maximum observed drug concentration (Cmax) | By week 3
Comparison of ELA026 Area under the curve plasma concentration versus time curve (AUC) | By week 3

CONTACTS AND LOCATIONS:
Locations (2):
- Celerion, Lincoln, Nebraska, United States
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No